CLINICAL TRIAL: NCT01777763
Title: Pharmacokinetics and Safety of Solid Oral Posaconazole (SCH 56592) in Subjects at High Risk for Invasive Fungal Infections (Phase 1b; Protocol No. P05615)
Brief Title: Pharmacokinetics and Safety of Posaconazole Tablet in Participants at High Risk for Invasive Fungal Infections (MK-5592-065/P05615)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P05615; 2008-006684-36 (EudraCT Number); 5592-065 (Other: Merck)
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Results first posted 2013-03-28 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Fungal Infections
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posaconazole 200 mg (Experimental): Posaconazole 200 mg (two 100 mg tablets) twice daily (BID) on Day 1 followed by 200 mg (two 100 mg tablets) once daily (QD) for up to 28 days
  Interventions: Drug: Posaconazole 200 mg
- Posaconazole 300 mg (Experimental): Posaconazole 300 mg (three 100 mg tablets) BID on Day 1 followed by 300 mg (three 100 mg tablets) QD for up to 28 days
  Interventions: Drug: Posaconazole 300 mg

INTERVENTIONS:
Drug: Posaconazole 200 mg
  Other Names: SCH 056592; MK-5592; Noxafil®
  Arms: Posaconazole 200 mg
Drug: Posaconazole 300 mg
  Other Names: SCH 056592; MK-5592; Noxafil®
  Arms: Posaconazole 300 mg

SUMMARY:
The purpose of this study is to collect pharmacokinetic (PK) information related to how well posaconazole tablet is distributed in the body and to determine the safety of this new formulation. The study consists of a Phase 1B study that includes participants with neutropenia undergoing chemotherapy for acute myelogenous leukemia (AML) or myelodysplasia (MDS) and a Phase 3 study that includes participants who are undergoing chemotherapy for AML or MDS and participants who are recipients of allogeneic hematopoietic stem cell transplant (HSCT).

DETAILED DESCRIPTION:
Participants with a blood disease or cancer that can affect their infection-fighting white blood cells and those who have undergone a hematopoietic stem cell transplant (HSCT) and are receiving immunosuppressive therapy and have or are at risk of graft-vs-host disease (GVHD) are eligible for the study. These blood diseases and their treatments can weaken the immune system and may put individuals at high risk for a serious fungal infection of their internal organs or blood (invasive fungal infection). As these infections can be hard to detect early and can be life-threatening, many physicians believe that individuals diagnosed with these diseases should receive antifungal therapy to try to lower their risk of getting this type of infection.

Enrollment into this study will take place in several stages (parts). The determination of which part a participant will be in is based on which part is open at the site at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >34 kg (75 lb) and of any race/ethnicity
* Able to swallow oral tablets whole
* Anticipated (likely to develop within 3-5 days) or documented neutropenia due to chemotherapy, chemotherapy for a new diagnosis of acute myelogenous leukemia (AML), or AML in first relapse; myelodysplastic syndromes (MDS) in transformation to AML; allogeneic hematopoietic stem cell transplant (HSCT) participants in the pre-engraftment period or in the post-engraftment period if they are receiving immunosuppressive therapy for graft versus host disease

Exclusion Criteria:

- Female must not be pregnant, must not intend to become pregnant

during the study, and must not be nursing

* History of hypersensitivity to azoles
* Moderate or severe liver dysfunction defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels greater than three times the upper limit of normal (ULN), AND a total bilirubin level greater than two times the ULN
* Electrocardiogram (ECG) with corrected QTc interval greater than 500 msec
* Posaconazole within 10 days before study enrollment
* Receipt of systemic antifungal therapy within 30 days of study enrollment for reasons other than antifungal prophylaxis
* Evidence of known or suspected invasive or systemic fungal infection at baseline
* Known or suspected history of Gilbert's disease
* Creatinine clearance levels below 30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Duarte RF, Lopez-Jimenez J, Cornely OA, Laverdiere M, Helfgott D, Haider S, Chandrasekar P, Langston A, Perfect J, Ma L, van Iersel ML, Connelly N, Kartsonis N, Waskin H. Phase 1b study of new posaconazole tablet for prevention of invasive fungal infections in high-risk patients with neutropenia. Antimicrob Agents Chemother. 2014 Oct;58(10):5758-65. doi: 10.1128/AAC.03050-14. Epub 2014 Jul 21. PMID 25049247
- [Result] Cornely OA, Duarte RF, Haider S, Chandrasakar P, Helfgott D, Lopez J, Candoni A, Raad I, Laverdiere M, Langston A, Van Iersel M, Connelly N, Waskin H. Phase 3 Pharmacokinetics and Safety Study of Posaconazole Tablet in Patients at Risk for Invasive Fungal Infection. J Antimicrob Chemother. 2015;[e-pub 26Nov2015]. doi: 10.1093/jac/dkv380
- [Derived] de Almeida C, Wong M, Kleijn HJ, Wrishko RE. Predicted Bezlotoxumab Exposure in Patients Who Have Received a Hematopoietic Stem Cell Transplant. Clin Ther. 2023 Apr;45(4):356-362. doi: 10.1016/j.clinthera.2023.02.006. Epub 2023 Mar 9. PMID 36906440
- [Derived] Cornely OA, Duarte RF, Haider S, Chandrasekar P, Helfgott D, Jimenez JL, Candoni A, Raad I, Laverdiere M, Langston A, Kartsonis N, Van Iersel M, Connelly N, Waskin H. Phase 3 pharmacokinetics and safety study of a posaconazole tablet formulation in patients at risk for invasive fungal disease. J Antimicrob Chemother. 2016 Mar;71(3):718-26. doi: 10.1093/jac/dkv380. Epub 2015 Nov 26. PMID 26612870

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Started | 20 | 210
Completed | 16 | 163
Not Completed | 4 | 47
Not completed — Adverse Event | 2 | 32
Not completed — Protocol Violation | 1 | 7
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Treatment Failure | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg | Total
Number analyzed (Participants) | 20 | 210 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.2) | 51.0 (14.1) | 51.0 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 79 | 87
  Male | 12 | 131 | 143

OUTCOME MEASURES:

1. Primary Outcome: Average Concentration (Cavg) of Posaconazole Tablet
Description: Posaconazole steady-state concentrations of posaconazole in the plasma reached after regular and repeated dosing were used to estimate pharmacokinetic (PK) parameters for each participant where Cavg was defined as area under the plasma concentration versus time curve divided by the dosing interval.
  Blood samples for the assessment of Cavg were collected on Day 1 and Day 8 predose and then at specified time points up to 24 hours postdose.
Time Frame: Predose on Day 1 up to 24 hours postdose on Day 8
Population: The Cavg PK population included participants who met the inclusion/exclusion criteria, complied with protocol procedures including collection of specified PK and dosing parameters, had no major protocol violations, and had documented adherence to dosing and PK regimens through the Day 8 steady-state visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Number analyzed (Participants) | 18 | 50
ng/mL | 981 (475) | 1580 (667)

2. Primary Outcome: Minimum Concentration (Cmin) of Posaconazole Tablet
Description: Cmin was defined as posaconazole trough level immediately before a participant received the dose of posaconazole tablets on the specified day. Trough (Cmin) level blood samples for determination of posaconazole in plasma were collected for all participants on Day 1, Day 2, Day 3, and Day 8. On Day 1, the trough level sample was collected the before the first dose of study drug. On Day 2, trough samples were collected approximately 12 hours after the second dose of study drug was administered on Day 1. On all subsequent days, trough samples were collected approximately 24 hours following the previous day's dose of study drug.
Time Frame: Predose on Day 1 up to 24 hours postdose on Day 8
Population: The Cmin PK population included participants who met the inclusion/exclusion criteria, complied with protocol procedures including collection of specified PK and dosing parameters, had no major protocol violations, and had documented adherence to dosing and PK regimens through the Day 8 steady-state visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Number analyzed (Participants) | 18 | 50
ng/mL | 812 (443) | 1310 (647)

3. Primary Outcome: Maximum Concentration (Cmax) of Posaconazole Tablet
Description: Blood samples for the assessment of Cmax were collected on Day 1 and Day 8 predose and then at specified time points up to 24 hours postdose.
Time Frame: Predose on Day 1 up to 24 hours postdose on Day 8
Population: The Cmax PK population included participants who met the inclusion/exclusion criteria, complied with protocol procedures including collection of specified PK and dosing parameters, had no major protocol violations, and had documented adherence to dosing and PK regimens through the Day 8 steady-state visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Number analyzed (Participants) | 18 | 50
ng/mL
  Day 1 | 652 (217) | 908 (354)
  Day 8 | 1310 (617) | 2090 (798)

4. Primary Outcome: Time to Maximum Concentration (Tmax) of Posaconazole Tablet
Description: Blood samples for the assessment of Tmax were collected on Day 1 and Day 8 predose and then at specified time points up to 24 hours postdose.
Time Frame: Predose on Day 1 up to 24 hours postdose on Day 8
Population: The Tmax PK population included participants who met the inclusion/exclusion criteria, complied with protocol procedures including collection of specified PK and dosing parameters, had no major protocol violations, and had documented adherence to dosing and PK regimens through the Day 8 steady-state visit.
Measure: Median (Full Range); unit: Hours
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Number analyzed (Participants) | 18 | 50
Hours
  Day 1 | 4 [1.9 to 4.1] | 4 [1.8 to 12.0]
  Day 8 | 4 [2.0 to 8.1] | 4 [1.3 to 8.3]

5. Primary Outcome: Apparent Total Body Clearance (CL/F) for Posaconazole Tablet
Description: Blood samples for the assessment of CL/F, the rate at which posaconazole was removed from the body, were collected on Day 1 and Day 8 predose and then at specified time points up to 24 hours postdose.
Time Frame: Predose on Day 1 up to 24 hours postdose on Day 8
Population: The CL/F PK population included participants who met the inclusion/exclusion criteria, complied with protocol procedures including collection of specified PK and dosing parameters, had no major protocol violations, and had documented adherence to dosing and PK regimens through predose on the Day 8 steady-state visit.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Number analyzed (Participants) | 18 | 50
L/hr | 10.9 (5.80) | 9.39 (4.20)

6. Other Pre Specified Outcome: Number of Participants Surviving at Day 65
Description: Number of Participants Alive at Day 65
Time Frame: Day 65
Population: The safety population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Number analyzed (Participants) | 20 | 210
Participants | 18 | 192

7. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: AEs are any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a study drug, whether or not considered related to this study drug. Treatment-emergent AEs are any events not present before starting study drug treatment or any events that were present before treatment that worsened in either intensity or frequency after exposure to study drug.
Time Frame: Up to Day 65
Population: The safety population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Number analyzed (Participants) | 20 | 210
Participants | 20 | 207

8. Other Pre Specified Outcome: Number of Participants With Treatment-Related AEs
Description: AEs are any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a study drug, whether or not considered related to this study drug. Treatment-related AEs were considered by the investigator to be related to the study drug.
Time Frame: Up to Day 65
Population: The safety population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Number analyzed (Participants) | 20 | 210
Participants | 10 | 84

9. Other Pre Specified Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: AEs are any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a study drug, whether or not considered related to this study drug. These AEs resulted in participants stopping study drug treatment. This measure includes participants who discontinued due to AEs and also includes treatment failures that were attributed to AEs.
Time Frame: Up to Day 28
Population: The safety population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Number analyzed (Participants) | 20 | 210
Participants | 3 | 38

ADVERSE EVENTS:
Time Frame: Up to Day 65
Arm/Group | Posaconazole 200 mg | Posaconazole 300 mg
Serious Adverse Events (participants affected / at risk) | 6/20 | 69/210
Other Adverse Events (participants affected / at risk) | 20/20 | 186/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole 200 mg (N=20) | Posaconazole 300 mg (N=210)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 11 (12)
MICROANGIOPATHIC HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
SPLENIC HAEMORRHAGE (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 0 (0) | 1 (1)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 4 (4)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
DISEASE PROGRESSION (General disorders) | 0 (0) | 1 (1)
DRUG INTERACTION (General disorders) | 0 (0) | 2 (2)
GENERALISED OEDEMA (General disorders) | 0 (0) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 0 (0) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 3 (4)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 0 (0) | 1 (1)
GRAFT VERSUS HOST DISEASE IN INTESTINE (Immune system disorders) | 0 (0) | 1 (1)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 3 (3)
CYTOMEGALOVIRUS VIRAEMIA (Infections and infestations) | 0 (0) | 2 (2)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
KLEBSIELLA INFECTION (Infections and infestations) | 0 (0) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION FUNGAL (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 2 (2)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA FUNGAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 0 (0) | 1 (1)
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 (0) | 2 (2)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 5 (6)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 2 (3)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ZYGOMYCOSIS (Infections and infestations) | 0 (0) | 1 (1)
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRANSPLANT FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 2 (2)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 3 (4)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 2 (2)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 1 (1)
WEIGHT INCREASED (Investigations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
POLYCYTHAEMIA VERA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
T-CELL PROLYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
SINUS HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole 200 mg (N=20) | Posaconazole 300 mg (N=210)
ANAEMIA (Blood and lymphatic system disorders) | 5 (13) | 22 (56)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 (5) | 34 (40)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (8) | 15 (19)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 7 (13) | 28 (72)
BRADYCARDIA (Cardiac disorders) | 2 (2) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 13 (19)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 9 (12)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (6) | 23 (26)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 14 (15)
CONSTIPATION (Gastrointestinal disorders) | 7 (7) | 20 (21)
DIARRHOEA (Gastrointestinal disorders) | 8 (8) | 59 (91)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 13 (13)
HAEMORRHOIDS (Gastrointestinal disorders) | 2 (2) | 11 (12)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 8 (11)
NAUSEA (Gastrointestinal disorders) | 4 (6) | 55 (65)
ORAL PAIN (Gastrointestinal disorders) | 3 (3) | 2 (2)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 1 (1)
VOMITING (Gastrointestinal disorders) | 8 (8) | 27 (33)
ASTHENIA (General disorders) | 6 (6) | 19 (19)
CATHETER SITE ERYTHEMA (General disorders) | 2 (2) | 20 (22)
CHEST PAIN (General disorders) | 3 (3) | 7 (7)
CHILLS (General disorders) | 6 (9) | 22 (28)
FATIGUE (General disorders) | 2 (2) | 14 (16)
MUCOSAL INFLAMMATION (General disorders) | 6 (9) | 29 (35)
OEDEMA PERIPHERAL (General disorders) | 2 (3) | 33 (39)
PYREXIA (General disorders) | 6 (8) | 57 (84)
CHOLESTASIS (Hepatobiliary disorders) | 2 (2) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 2 (3) | 3 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 15 (22)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 12 (14)
HAEMOGLOBIN DECREASED (Investigations) | 2 (3) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (4) | 17 (18)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 13 (13)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (4) | 46 (56)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2) | 20 (24)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 4 (5) | 17 (19)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 13 (13)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (12)
DIZZINESS (Nervous system disorders) | 0 (0) | 13 (14)
HEADACHE (Nervous system disorders) | 4 (4) | 30 (36)
ANXIETY (Psychiatric disorders) | 0 (0) | 14 (14)
INSOMNIA (Psychiatric disorders) | 3 (3) | 15 (16)
DYSURIA (Renal and urinary disorders) | 1 (1) | 11 (12)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 35 (37)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 17 (17)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 30 (43)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (13)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 12 (14)
PETECHIAE (Skin and subcutaneous tissue disorders) | 2 (2) | 19 (22)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 16 (17)
RASH (Skin and subcutaneous tissue disorders) | 5 (5) | 34 (39)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
HYPERTENSION (Vascular disorders) | 3 (3) | 23 (24)
HYPOTENSION (Vascular disorders) | 3 (4) | 12 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.